CLINICAL TRIAL: NCT04357366
Title: suPAR-guided Anakinra Treatment for Validation of the Risk and Early Management of Severe Respiratory Failure by COVID-19: The SAVE Open-label, Non-randomized Single-arm Trial
Brief Title: suPAR-guided Anakinra Treatment for Validation of the Risk and Management of Respiratory Failure by COVID-19 (SAVE)
Acronym: SAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SAVE; 2020-001466-11 (EudraCT Number)
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Virus Diseases; Corona Virus Infection; Lower Respiratory Tract Infection Viral
Keywords: COVID-19; SARS-CoV-2; Anakinra; suPAR
MeSH Terms: conditions — COVID-19; Virus Diseases; Coronavirus Infections | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Treatment with anakinra
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anakinra (Experimental): Patients will receive 100mg of anakinra subcutaneously once daily for ten days. The drugs should be administered on the same time ± 2 hours every day. All other administered drugs are allowed. In case the patient is discharged home before the completion of 10 days of treatment, it is at the discretion of the investigator to suggest treatment continuation at home. In case such a decision is taken, the patient will be provided the required number of pre-filled syringes for daily self-injection. In this case, the patient should return the empty used syringes within 30 days.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Treatment with 100mg Anakinra subcutaneously (sc) once daily for ten days
  Other Names: Kineret

SUMMARY:
In the SAVE study patients with lower respiratory tract infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at high risk for progression to serious respiratory failure will be detected using the suPAR biomarker. They will begin early treatment with anakinra in the effort to prevent progression in serious respiratory failure.

DETAILED DESCRIPTION:
The major hurdle of Coronavirus disease 2019 (COVID-19) is the early recognition of the patients at high risk for the development of severe respiratory failure (SRF). If this can be achieved early, then appropriate immunomodulatory treatment may be administered to prevent development of SRF. This scenario is extremely visionary since it prevents the development of the major fatal consequence of COVID-19 but also alleviates the heavy medical and financial burden of Intensive Care Unit (ICU) admission.

Current evidence suggests that SARS-CoV-2 activates endothelial function which leads to over-production of D-dimers. Urokinase plasminogen activator receptor (uPAR) is anchored to the cell membranes of the lung endothelial cells. As result of the activation of kallikrein, uPAR is cleaved and enters the systemic circulation as the soluble counterpart suPAR. Preliminary unpublished data from 57 Greek patients hospitalized after March 1st, 2020 in Greek hospitals due to pneumonia by confirmed SARS-CoV-2 infection showed that those with suPAR admission levels ≥ 6 ng/ml had greater risk for the development of SRF within 14 days than patients with suPAR less than 6ng/ml. The sensitivity of suPAR to detect these patients was 85.9% and the positive predictive value 85.9%. It needs to be underlined that all 21 Greek patients with suPAR≥ 6ng/ml were under treatment with hydroxychloroquine and azithromycin. These data were confirmed in 15 patients hospitalized for pneumonia by SARS-CoV-2 in Rush Medical Center at Chicago.

This prognostic ability of suPAR for unfavourable outcome is not presented for the first time; in the TRIAGE III trial that was conducted among 4,420 admissions in the emergency department in Denmark the interquartile range of suPAR was between 2.6 and 4.7 ng/ml in 30-day survivors and between 6.7 and 11.8 ng/ml in 30-day non-survivors. Previous data from the Hellenic Sepsis Study Group on 1,914 patients clearly shows a high prognostic utility of admission suPAR for 28-day mortality.

It is obvious that suPAR can early identify the start of such a type of inflammatory process in the lung parenchyma that has will soon be intensified. A recent publication has shown that this is due to the early release of interleukin-1α (IL-1α) from lung epithelial cells that are infected by the virus. This IL-1α acts as a promoting factor that stimulates the production of IL-1β and of a further cytokine storm from alveolar macrophages.

Anakinra is the only marketed product that inhibits both IL-1β and IL-1α and hence it is able to block an inflammatory response early on and to prevent the downstream inflammatory cascade. suPAR can be used as the biomarker tool to indicate patients with COVID-19 pneumonia in risk of SRF and for whom early start of anakinra may prevent development of SRF.

Anakinra is a safe drug that has been licensed for chronic subcutaneous administration in rheumatoid arthritis, refractory gout and chronic auto-inflammatory disorders. The safety profile was further proven when it was administered in two randomized clinical trials where more than 1,500 critically ill patients with severe sepsis were intravenously treated.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Male or female gender
* In case of women, unwillingness to remain pregnant during the study period.
* Written informed consent provided by the patient or by one first-degree relative/spouse in case of patients unable to consent
* Confirmed infection by SARS-CoV-2 virus using molecular techniques as defined by the World Health Organization
* Findings in chest-X-ray or in chest computed tomography compatible with lower respiratory tract infection
* Plasma suPAR ≥6ng/ml

Exclusion Criteria:

* Age below 18 years
* Denial for written informed consent
* Any stage IV malignancy
* Any do not resuscitate decision
* Any primary immunodeficiency
* Less than 1,500 neutrophils/mm3
* Known hypersensitivity to anakinra
* Oral or IV intake of corticosteroids at a daily dose equal or greater than 0.4 mg prednisone for a greater period than the last 15 days.
* Any anti-cytokine biological treatment the last one month
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Severe hepatic failure
* Severe renal failure
* Any need for CPAP or mechanical ventilation
* Any pO2/FiO2 ratio less than 150

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
The ratio of patients who will develop serious respiratory failure (SRF) | Visit study day 14
  The primary study endpoint is the ratio of patients who will develop serious respiratory failure SRF until day 14. Patients dying before study visit of day 14 are considered achieving the primary endpoint.

SECONDARY OUTCOMES:
Comparison of the rate of patients who will develop serious respiratory failure (SRF) until day 14 with comparators from Hellenic Sepsis Study Group Database receiving standard-of-care treatment | Visit study day 14
  Evaluation of clinical data (pO2/FiO2 and need of mechanical ventilation) between baseline and study visit day 14 will be compared with comparators from Hellenic Sepsis Study Group Database
Change of scoring for respiratory symptoms in enrolled subjects between days 1 and 7 | Visit study day 1, visit study day 7
  Change of scoring for respiratory symptoms (evaluation of cough, chest pain, shortness of breath and sputum) in enrolled subjects between days 1 and 7
Change of scoring for respiratory symptoms in enrolled subjects between days 1 and 14 | Visit study day 1, visit study day 14
  Change of scoring for respiratory symptoms (evaluation of cough, chest pain, shortness of breath and sputum) in enrolled subjects between days 1 and 14
Change of SOFA score in enrolled subjects between days 1 and 7 | Visit study day 1, visit study day 7
  Change of Sequential organ failure assessment (SOFA) score of enrolled subjects between days 1 and 7 (Sequential organ failure assessment range 0-24, high score associated with worst outcome)
Change of Sequential organ failure assessment (SOFA) score in enrolled subjects between days 1 and 14 | Visit study day 1, visit study day 14
  Change of Sequential organ failure assessment (SOFA) score of enrolled subjects between days 1 and 14 (Sequential organ failure assessment range 0-24, high score associated with worst outcome)
Change of peripheral mononuclear blood cells' (PBMCs) functionality between days 1 and 7 | Visit study day 1, visit study day 7
  Change of peripheral mononuclear blood cells' (PBMCs) functionality of enrolled subjects will be compared between days 1 and 7
Change of plasma inflammatory mediators levels between days 1 and 7 | Visit study day 1, visit study day 7
  Change of plasma inflammatory mediators measured levels will be compared between days 1 and 7
Rate of Mortality | Visit study day 30
  Mortality on day 30
Rate of Mortality | Visit study day 90
  Mortality on day 90
Change of gene expression between days 1 nad 7 | days 1 and 7
  Transcriptional, proteomic and metabolomic change will be compared between days 1 and 7
Safety of anakinra | Last patients visit, Day 90
  Safety of anakinra
Association between the time interval from hospital admission until start of anakinra and the incidence of SRF | Visit day 14
  Association between the time interval from hospital admission until start of anakinra and the incidence of SRF
Correlation between time interval and the occurrence of SAA under treatment with anakinra | Visit day 14
  Correlation between time interval and the occurrence of SAA under treatment with anakinra
Association between radiological opacities in chest computed tomography and the incidence of SRF under anakinra treatment | Visit day 14
  Association between radiological opacities in chest computed tomography and the incidence of SRF under anakinra treatment
Association of the efficacy of anakinra for subgroups of patients; the studied subgroups will be the quartiles of the respiratory ratio (pO2/FiO2) at admission; the main comorbidities; the WHO classification | Visit day 14
  Association of the efficacy of anakinra for subgroups of patients; the studied subgroups will be the quartiles of the respiratory ratio (pO2/FiO2) at admission; the main comorbidities; the WHO classification

CONTACTS AND LOCATIONS:
Overall Officials: Simeon Metallidis, MD, PhD, Principal Investigator — Aristotle University of Thessaloniki, Medical School
Locations (28):
- Greece (28):
  - COVID-19 Department, General Hospital of Attica SISMANOGLEIO-AMALIA FLEMING, Marousi, Athens
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - Department of Internal Medicine, I PAMMAKARISTOS Hospital, Athens
  - 1st Department of InternalMedicine, General Hospital of Athens KORGIALENIO-BENAKIO E.E.S., Athens
  - 1st Department of Internal Medicine, General Hospital of Athens G. GENNIMATAS, Athens
  - 1st University Department of Internal Medicine, General Hospital of Athens LAIKO, Athens
  - 1st University Departmentof Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseasesof Athens, Athens
  - 2nd University Department of Internal Medicine, IPPOKRATEION General Hospital of Athens, Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens I SOTIRIA, Athens
  - Department of Internal Medicine, General Hospital of Chest Diseases of Athens I SOTIRIA, Athens
  - Department of Clinical Therapeutics, ALEXANDRA General Hospital of Athens, Athens
  - 1st Department of Internal Medicine Amalia Fleming General Hospital, Athens
  - 1st Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 1st Department of Internal Medicine, General Hospital of Nea Ionia CONSTANTOPOULIO-PATISION, Athens
  - 1st Department of Internal Medicine, General Hospital of Voula ASKLEPIEIO, Athens
  - 2nd Department of Internal Medicine, 251 Air Force General Hospital, Athens
  - 2nd Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 3rd Department of Internal Medicine, General Hospital of Athens KORGIALENEIO-BENAKEIO E.E.S., Athens
  - 5th Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - Department of Internal Medicine, General Hospital of Athens ELPIS, Athens
  - Department of Infectious Diseases, General Hospital of Kerkira, Corfu
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Ioannina
  - Department of Internal Medicine, General Hospital of Katerini, Katerini
  - Department of Internal Medicine, University General Hospital of Larissa, Larissa
  - Department of Internal Medicine, General Hospital of Larisa KOUTLIMBANEIO & ΤΡΙΑΝΤΑFΥLLΕΙΟ, Larissa
  - Department of Internal Medicine, University General Hospital of Patras PANAGIA I VOITHIA, Pátrai
  - 2nd Department of Internal Medicine, General Hospital of Piraeus TZANEIO, Piraeus
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kyriazopoulou E, Akinosoglou K, Florou E, Kouriannidi E, Bogosian A, Tsachouridou O, Syrigos KN, Gatselis N, Milionis H, Papanikolaou IC, Sympardi S, Dafni M, Alevizou A, Amvrazi AV, Alexandrou E, Archontoulis K, Argyraki K, Alexiou Z, Georgiou Y, Gkogka D, Kyrailidi F, Kalyva V, Nikolopoulou T, Ioannou S, Bakakos P, Karathanassiou G, Koklanos K, Miletis DN, Tili AM, Vakkas L, Vila I, Panagopoulos P, Samarkos M, Chrysos G, Dalekos GN, Poulakou G, Metallidis S, Giamarellos-Bourboulis EJ. Anakinra efficacy in COVID-19 pneumonia guided by soluble urokinase plasminogen activator receptor: Association with the inflammatory burden of the host. Int J Antimicrob Agents. 2025 Jan;65(1):107405. doi: 10.1016/j.ijantimicag.2024.107405. Epub 2024 Dec 6. PMID 39647797
- [Derived] Kyriazopoulou E, Dalekos GN, Metallidis S, Poulakou G, Papanikolaou IC, Tzavara V, Argyraki K, Alexiou Z, Panagopoulos P, Samarkos M, Chrysos G, Tseliou A, Milionis H, Sympardi S, Vasishta A, Giamarellos-Bourboulis EJ. HEPARIN-BINDING PROTEIN LEVELS PREDICT UNFAVORABLE OUTCOME IN COVID-19 PNEUMONIA: A POST HOC ANALYSIS OF THE SAVE TRIAL. Shock. 2024 Mar 1;61(3):395-399. doi: 10.1097/SHK.0000000000002315. Epub 2024 Jan 19. PMID 38517242
- [Derived] Keur N, Saridaki M, Ricano-Ponce I, Netea MG, Giamarellos-Bourboulis EJ, Kumar V. Analysis of inflammatory protein profiles in the circulation of COVID-19 patients identifies patients with severe disease phenotypes. Respir Med. 2023 Oct;217:107331. doi: 10.1016/j.rmed.2023.107331. Epub 2023 Jun 25. PMID 37364721
- [Derived] Samaras C, Kyriazopoulou E, Poulakou G, Reiner E, Kosmidou M, Karanika I, Petrakis V, Adamis G, Gatselis NK, Fragkou A, Rapti A, Taddei E, Kalomenidis I, Chrysos G, Bertoli G, Kainis I, Alexiou Z, Castelli F, Saverio Serino F, Bakakos P, Nicastri E, Tzavara V, Kostis E, Dagna L, Koukidou S, Tzatzagou G, Chini M, Bassetti M, Trakatelli C, Tsoukalas G, Selmi C, Samarkos M, Pyrpasopoulou A, Masgala A, Antonakis E, Argyraki A, Akinosoglou K, Sympardi S, Panagopoulos P, Milionis H, Metallidis S, Syrigos KN, Angel A, Dalekos GN, Netea MG, Giamarellos-Bourboulis EJ. Interferon gamma-induced protein 10 (IP-10) for the early prognosis of the risk for severe respiratory failure and death in COVID-19 pneumonia. Cytokine. 2023 Feb;162:156111. doi: 10.1016/j.cyto.2022.156111. Epub 2022 Dec 14. PMID 36529030
- [Derived] Renieris G, Karakike E, Gkavogianni T, Droggiti DE, Stylianakis E, Andriopoulou T, Spanou VM, Kafousopoulos D, Netea MG, Eugen-Olsen J, Simard J, Giamarellos-Bourboulis EJ. IL-1 Mediates Tissue-Specific Inflammation and Severe Respiratory Failure in COVID-19. J Innate Immun. 2022;14(6):643-656. doi: 10.1159/000524560. Epub 2022 May 11. PMID 35545011
- [Derived] Kyriazopoulou E, Panagopoulos P, Metallidis S, Dalekos GN, Poulakou G, Gatselis N, Karakike E, Saridaki M, Loli G, Stefos A, Prasianaki D, Georgiadou S, Tsachouridou O, Petrakis V, Tsiakos K, Kosmidou M, Lygoura V, Dareioti M, Milionis H, Papanikolaou IC, Akinosoglou K, Myrodia DM, Gravvani A, Stamou A, Gkavogianni T, Katrini K, Marantos T, Trontzas IP, Syrigos K, Chatzis L, Chatzis S, Vechlidis N, Avgoustou C, Chalvatzis S, Kyprianou M, van der Meer JW, Eugen-Olsen J, Netea MG, Giamarellos-Bourboulis EJ. An open label trial of anakinra to prevent respiratory failure in COVID-19. Elife. 2021 Mar 8;10:e66125. doi: 10.7554/eLife.66125. PMID 33682678